CLINICAL TRIAL: NCT00760110
Title: Usefulness of Home Blood Pressure Measurement in the Morning in Type 2 Diabetic Patients: Long-Term Results of a Prospective Longitudinal Study
Brief Title: A Cohort Study of Morning Home Blood Pressure Measurement in Type 2 Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Nagaoka Red Cross Hospital (Other)
Responsible Party: Kyuzi Kamoi, Nagaoka Red Cross Hospital
Other Study IDs: 1
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Hypertension; Type 2 Diabetes
Keywords: Morning BP; Clinic BP; micro- and macrovascular complications
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 Morning hypertension and normotension: Based on HBP, subjects were divided into MH and MN patients
  Interventions: Device: blood pressure measurements based on HBP or CBP
- 2 Clinic hypertension and normotension: Based on CBP, subjects were divided into CH and CN patients
  Interventions: Device: blood pressure measurements based on HBP or CBP

INTERVENTIONS:
Device: blood pressure measurements based on HBP or CBP — To clarify which of HBP or CBP provides the stronger predictive power for the outcomes, the 400 patients were classified as with or without hypertension based on HBP and CBP measurements at baseline

SUMMARY:
Previous cross-sectional studies have demonstrated that blood pressure (BP) measurements at home (HBP) in the morning offer stronger predictive power for micro- and macrovascular complications in patients with type 1 and 2 diabetes than casual/clinic blood pressure measurements (CBP). The present study examined which of HBP or CBP provides the stronger predictive power for outcomes by comparing cumulative events between hypertensive and normotensive patients over 6 years in a prospective, longitudinal study of patients with type 2 diabetes.

DETAILED DESCRIPTION:
RESEARCH DESIGN AND METHODS

１.Subjects. After a detailed baseline examination, 400 Japanese subjects were followed up for all-cause mortality and morbidity. All participants visited our clinic regularly. Mean survey duration of all patients was 42.1±20.0 months (range, 3-72 months).Type 2 diabetes was diagnosed according to World Health Organization criteria.At the beginning of the study, 329 patients(82%)were receiving treatment with oral hypoglycemic drugs and/or insulin regimens for diabetes mellitus and 196 patients (49%) were receiving treatment with various anti-hypertensive drugs (angiotensin-converting enzyme inhibitors, angiotensin receptor blockers, calcium channel blocker and others) for hypertension. Mean disease duration was 13±8 years (range, 0-40 years). Mean values for other baseline measurements were as follows: BMI,23.7±3.4 kg/m2;HbA1c,6.7±1.1%; triglycerides,150±112 mg/dl;total cholesterol,198±32 mg/dl; LDL,110±29 mg/dl; and HDL,60±19 mg/dl.All patients were fully informed about the purposes and procedures for the study and provided oral consent at enrolment.

2. Baseline and follow-up assessment. Participants were examined using the same methods reported previously (1,2). Briefly, all chemical laboratory data were obtained at each visit without fasting in the morning. BP was measured in the clinic and at home on waking in the morning. Clinic hypertension (CH) and morning hypertension (MH) were defined as systolic BP (SBP)>=130 mmHg and/or diastolic BP (DBP)>=85 mmHg, while clinic normotension (CN) and morning normotension (MN) were defined as SBP <130 mmHg and DBP <86 mmHg, respectively. Microalbuminuria and clinical albuminuria were defined as urinary albumin excretion rate >=30 mg/g creatinine and >=300 mg/g creatinine, respectively.

Microvascular complications were checked for at baseline and every 3 to 6 months throughout the study. Severity of nephropathy was determined using 4 categories: normal; microalbuminuria; clinical albuminuria; and dialysis. Severity of retinopathy was categorized as: normal; non-proliferative retinopathy; pre-proliferative retinopathy; and proliferative retinopathy. Development of changing microvascular events defined according to a change of at least 1 step from baseline (3,4). Macrovascular complications were coronary heart disease (CHD) and cerebrovascular disease (CVD). These events were confirmed by medical history, including contents of treatment. New or worsened (recurrent) events were defined based on clinical manifestations and treatment throughout the study.

At baseline, HT or NTs were determined on the basis of HBP and CBP measurements. Based on HBP, subjects were divided into MH and MN patients, and each endpoint was determined within the survey duration, as defined by the patient displaying sustenance of the same BP status. That is, survey duration varied between individual patients and was defined as the period of time until an MH patient at baseline displayed a change to MN, or until an MN patient at baseline displayed a change to MH. Mean survey duration until endpoints was 29.5±21.1 months(range, 3-72 months).

Also, based on CBP, subjects were divided into CH and CN patients. These patients were followed using the same methods used for MH and MN. Mean survey duration until endpoints was 34.9±22.3 months (range,3-72 months), which was significantly longer than that based on HBP (P<0.001).

For ethical reasons, patients were treated with various anti-hypertensive, anti-diabetic, anti-dyslipidemia and/or anti-hypercoagulation agents during the course of the study by the patients'own doctors as a part of continuing standard medical care.

3. Study endpoints and outcome measures. The primary endpoint was death from any cause. Secondary endpoints were new, worsened or improved microvascular events and new or worsened macrovascular events.

4. Statistical analysis

1. Baseline. Mean values were compared using Student's paired or unpaired t test. To compare the prevalence of micro- and macrovascular complications or medical treatment in patients with and without hypertension on the basis of HBP or CBP, Fischer's exact test with two-tailed P values was used, and then odds ratio and 95% confidence interval (CI) were calculated. If prevalence of an event was zero, 0.5 was added to all values before calculating the odds ratio and 95% CI.
2. Endpoints and outcome measures. Differences in outcomes for each endpoint of death and new or worsened micro- and macrovascular complications between sustained hypertensive and normotensive patients on the basis of HBP or CBP were assessed using survival curves calculated according to Kaplan-Meier methods, then compared by hazard ratio using the log-rank test. Within the survey time defined above, a time until censoring or death (or occurrence of the event) was calculated for each endpoint.
3. Risk factor assessment for outcomes. Risk factors related to outcomes determined statistically by log-rank test were assessed using hazard ratios by Cox proportional hazards model. For outcomes of microvascular complications, risk factors were determined in new, worsened or improved events. Omnibus tests were used to determine the appropriateness of Cox proportional hazards modeling. Confounding factors used in this analysis were variables with MH or CH at baseline and additional therapy for each disease.

Analysis was performed using Prism version 5.01 software (GraphPad Software, CA, USA) and the Dr. SPSSII for Windows (SPSS Japan, Tokyo, Japan). Two-tailed values of P<0.05 were defined as statistically significant.

References

1. Kamoi K, et al. Usefulness of home blood pressure measurement in the morning in type 2 diabetic patients. Diabetes Care 25:2218-2223, 2002
2. Kamoi K, et al.Usefulness of home blood pressure measurement in the morning in type 1 diabetic patients. Diabetes Care 26:2218-2223, 2003
3. The Diabetes Control and Complications Trial Research Group: The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med 329:977-986, 1993
4. Ohkubo Y, et al Intensive insulin therapy prevents the progression of diabetic microvascular complications in Japanese patients with non-insulin-dependent diabetes mellitus: a randomized prospective 6-year study. Diabetes Res Clin Pract 28:103-117, 1995

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with HBP and CBP measurements

Exclusion Criteria:

* Type 1 or 2 diabetic patients without HBP and CBP measurements

Ages: 23 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects comprised 400 Japanese patients with type 2 diabetes enrolled between 1999 and 2005.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 1997-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Death | Duration varied between individual patients and was as the period of time until MH or CH patient at baseline displayed a change to MN or CN, or until MN or CN patient at baseline displayed a change to MH or CH, respectively

SECONDARY OUTCOMES:
Microvascular complications | Duration varied between individual patients and was as the period of time until MH or CH patient at baseline displayed a change to MN or CN, or until MN or CN patient at baseline displayed a change to MH or CH, respectively
Macrovascular complications | Duration varied between individual patients and was as the period of time until MH or CH patient at baseline displayed a change to MN or CN, or until MN or CN patient at baseline displayed a change to MH or CH, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Kyuzi Kamoi, MD, Principal Investigator — Nagaoka Red Cross Hospital

REFERENCES:
- [Derived] Kamoi K, Ito T, Miyakoshi M, Minagawa S. Usefulness of home blood pressure measurement in the morning in patients with type 2 diabetes: long-term results of a prospective longitudinal study. Clin Exp Hypertens. 2010 May;32(3):184-92. doi: 10.3109/10641960903254513. PMID 20504126